CLINICAL TRIAL: NCT01546168
Title: Esophageal Deviation in Atrial Fibrillation Ablation: A Randomized Control Trial
Brief Title: Deviating the Esophagus in Atrial Fibrillation Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis: no statistically significant difference in the 2 study arms.
Sponsor: Vivek Reddy (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 11-0909
Record Dates: First submitted 2012-02-13; First posted 2012-03-07 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Deviation; Atrial Fibrillation; Ablation
Keywords: Atrial Fibrillation ablation; Esophageal Deviation; AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esophageal deviation (Experimental): esophageal deviation with IDE device during AF ablation
  Interventions: Device: esophageal deviation with IDE device
- temperature monitoring (No Intervention): luminal esophageal temperature monitoring, standard temperature monitoring alone

INTERVENTIONS:
Device: esophageal deviation with IDE device — esophageal deviation during AF ablation
  Arms: esophageal deviation

SUMMARY:
In this randomized double-blind study, the investigators would like to compare standard practice (i.e., use of luminal esophageal temperature monitoring) to that of esophageal deviation during AF ablation. The investigators hypothesize that the strategy of esophageal deviation will result in safer ablation strategy with a reduction in the incidence of esophageal injury as assessed by endoscopy.

DETAILED DESCRIPTION:
Catheter ablation is a commonly performed strategy employed for the treatment of atrial fibrillation. However ablation in the posterior wall of the left atrium can cause thermal injury to the esophagus. When significant thermal injury to the esophagus occurs, two significant complications can occur: 1) the formation of an atrio-esophageal fistula, and 2) gastrointestinal dysmotility. While the former is rate, it is an important complication since it can be fatal. The frequency of the latter complication is less well appreciated, but probably occurs in the range of 1:100 to 1:500. Currently luminal esophageal temperature monitoring is the most commonly employed modality to prevent such injury. However, there are limitations to its use, and atrio-esophageal fistulas have been reported even when using esophageal temperature monitoring. Esophageal deviation using either a TEE or EGD probe has been described in the literature, but the effectiveness and practicality of these techniques are suboptimal, and have therefore precluded their use in routine clinical practice. Recently, we have demonstrated that esophageal deviation is indeed possible using off-the-shelf equipment (a soft thoracic tube and endotracheal stylet) in patients undergoing AF ablation. In this randomized double-blind study, we will compare standard practice (i.e., use of luminal esophageal temperature monitoring) to esophageal deviation during AF ablation. We hypothesize that the strategy of esophageal deviation will result in safer ablation strategy with a reduction in the incidence of esophageal injury as assessed by endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 - Age < 80 yr
* Documentation of atrial fibrillation (AF)
* Referred for a first ever ablation procedure for AF (prior ablation of right-sided Typical flutter, or "limited" left-sided of an accessory pathway are permitted)
* General anesthesia
* All patients must understand and adhere to the requirements of the study and be willing to comply with the post study follow-up requirements.

Exclusion Criteria:

* Any reversible cause of AF (post-surgery, thyroid disorder, etc.)
* INR > 4.0 at the time of the procedure
* H/o of severe esophageal ulcers, strictures, esophagitis or GERD
* H/o Esophageal Surgery
* Prior surgical or catheter ablation procedure for AF (except right atrial flutter ablation)
* Any evidence of esophageal diverticulum or other structural abnormalities of the esophagus seen during baseline barium esophagogram
* Significant abnormality on Swallowing Impairment Score
* Mental impairment precluding signing consent or completing follow up
* Patients with any other significant uncontrolled or unstable medical condition
* Women who are known to be pregnant or have had a positive β-HCG test 7 days prior to procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Florida Hospital, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Texas Cardiac Arrhythmia Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November 2011, with enrollment beginning February 2012
Pre-assignment Details: 88 participants were consented, but 2 withdrew prior to randomization
Groups:
- Temperature Monitoring: luminal esophageal standing temperature monitoring alone
Period: Overall Study
Arm/Group | Esophageal Deviation | Temperature Monitoring
Started | 55 | 33
Completed | 51 | 33
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — ineligible after signing consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Esophageal Deviation | Temperature Monitoring | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.3) | 62.6 (8.6) | 61.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 24 | 27 | 51
Persistent AF [Count of Participants; unit: Participants] | 16 | 15 | 31
Paroxysmal AF [Count of Participants; unit: Participants] | 20 | 18 | 38
CHADS Score [Mean (Standard Deviation); unit: units on a scale] — CHADS score for Stroke Risk Assessment in Atrial Fibrillation CHADS is a mnemonic for Congestive Heart Failure, Hypertension, Age over 75 years, Diabetes Mellitus, and Stroke or TIA history CHADS Score >2 (CVA risk >5% per year) CHADS Score 1 (CVA risk >4% per year) CHADS Score 0 (low risk)
  units on a scale | 0.7 (0.8) | 1 (0.9) | 0.83 (0.9)
History of GERD [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Esophageal Injury
Description: The presence of esophageal injury as assessed by upper gastrointestinal endoscopy that is performed within 1 week of the procedure.
Time Frame: within 1 week of AF ablation procedure
Population: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Deviation | Temperature Monitoring
Number analyzed (Participants) | 36 | 33
Participants | 5 | 4

2. Secondary Outcome: Procedure Time
Description: Procedure time and fluoroscopic imaging with barium contrast time
Time Frame: day 1, duration ofAF ablation procedure
Population: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Esophageal Deviation | Temperature Monitoring
Number analyzed (Participants) | 36 | 33
minutes
  Fluoroscopy time | 21.1 (9.9) | 20.9 (18.3)
  Procedure duration | 3.39 (1.00) | 4.11 (1.07)

3. Secondary Outcome: Temperature
Description: Extent of temperature rise on the temperature monitoring probe
Time Frame: during AF ablation procedure (intraoperative)
Population: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Esophageal Deviation | Temperature Monitoring
Number analyzed (Participants) | 36 | 33
Celsius | 0.26 (0.2) | 1.1 (0.7)

4. Secondary Outcome: Swallowing Impairment Score
Description: Swallowing impairment during procedure - Scale from 0 (no impairment) to 4 (severe impairment).
Time Frame: during AF ablation procedure (intraoperative)
Population: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Esophageal Deviation | Temperature Monitoring
Number analyzed (Participants) | 36 | 33
units on a scale | 0.67 [0 to 4] | 0.27 [0 to 4]

ADVERSE EVENTS:
Description: 17 roll-in patients and two pre-procedure withdrawals are removed from the analysis.
Arm/Group | Esophageal Deviation | Temperature Monitoring
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/36 | 3/33
Other Adverse Events (participants affected / at risk) | 7/36 | 4/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esophageal Deviation (N=36) | Temperature Monitoring (N=33)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 2
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esophageal Deviation (N=36) | Temperature Monitoring (N=33)
Atrial Flutter (Cardiac disorders) | 3 | 0
Groin Hematoma (Renal and urinary disorders) | 1 | 0
Nausea with abdominal pain (Gastrointestinal disorders) | 2 | 1
Venous Thrombophlebitis (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes